CLINICAL TRIAL: NCT01477203
Title: Multimodal Assessment of Neurobiological Markers for Psychiatric Disorders
Acronym: MAN-BIOPSY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof.PD.Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FA103FC001; 2011-004860-31 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Major Depressive Disorder (MDD); Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Escitalopram (Active Comparator): 50 Major Depressive Disorder Patients and 50 Anxiety Disorder Patients will receive Escitalopram as medication
  Interventions: Drug: Escitalopram
- Remitted Patients (No Intervention)
- Healthy Controls (No Intervention)

INTERVENTIONS:
Drug: Escitalopram — 2-4 weeks, 5-10mg, max 20mg
  Arms: Escitalopram

SUMMARY:
MAN-BIOPSY pursues the concrete research question whether novel biological and psycho-physiological clusters or categories can be defined to improve treatment and minimize side effects in psychiatry, based on a synopsis of physiological, behavioural, genetic and endocrinological parameters. One major aspect of our research approach is its focuses on the identification of dysfunctions in fundamental information processing mechanisms and neurocomputational mechanisms, and is not restricted to symptom-oriented tasks.

The main objectives of MAN-BIOPSY are therefore

* to identify biological and psycho-physiological parameters for major depressive disorders and anxiety disorders, and
* to identify predictive markers for treatment response and type/severity of side effects for these disorders.

ELIGIBILITY:
Inclusion Criteria for patients:

* DSM-IV-TR diagnosis of MDD or an anxiety disorder (excluding PTSD, specific phobias, and bipolar disorder) by a structured clinical interview (SCID)
* aged 18 to 50 years
* drug-free within the last three months prior inclusion
* willingness and competence to sign the informed consent form

Inclusion Criteria for remitted subjects:

* a previous DSM-IV-TR diagnosis of MDD or an anxiety disorder (excluding PTSD, specific phobias, and bipolar disorder) but no symptoms at present, determined by SCID
* aged 18-50 years
* drug-free within the last three months prior inclusion
* willingness and competence to sign the informed consent form

Inclusion Criteria for healthy control subjects:

* Inclusion criteria for healthy control subjects are
* willingness and competence to sign the informed consent form
* aged 18-50 years
* drug-free

Exclusion Criteria:

* concomitant major internal or neurological illness
* concomitant psychiatric disorders (except depression and anxiety for patients, excluding PTSD, claustrophobia and bipolar disorder)
* ingestion of any antipsychotic, antidepressant, or anti-anxiety agent within the last three months prior to the screening visit
* current substance abuse
* failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 289 (Actual)
Dates: Start 2011-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
SSRI induced changes in BOLD (blood oxygen level dependent) response over time | 4 vears
SSRI induced changes in ERPs (event-related potentials) over time | 4 years

SECONDARY OUTCOMES:
biochemical data | 4 years
  these include steroid hormone levels, vitamins, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department for Psychiatrie and Psychotherapie, Vienna, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.meduniwien.ac.at/neuroimaging/
- See also: Related Info — http://biol-psy.univie.ac.at/